CLINICAL TRIAL: NCT00973492
Title: Impact of Functional Insulinotherapy on Blood Glucose Variability Indicators in Patients With Type 1 Diabetes
Acronym: VARIAFIT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Association Grenobloise pour le Developpement D'etudes et de Recherches en Physiopathologie Endocrinienne, Diabetologie et Maladies de la Nutrition (Other)
Responsible Party: Pr Pierre-Yves Benhamou, University Hospital Grenoble
Other Study IDs: 2007-A00903-50
Record Dates: First submitted 2009-09-07; First posted 2009-09-09 (Estimated); Last update posted 2009-09-09 (Estimated); Status verified 2009-09

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; functional insulinotherapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with functional insulinotherapy: There is only one group in this study. The participants will attend a functional insulinotherapy class.
  Interventions: Other: functional insulinotherapy class

INTERVENTIONS:
Other: functional insulinotherapy class — The functional insulinotherapy class lasts for 4 days. It is taught by 2 nurses, 2 dieticians and 2 physicians to 6 to 10 patients.
  On day 1, patients describe their difficulties with diabetes. Fast-acting insulin scales are elaborated from preprandial and postprandial blood glucose levels. At dinner, patients start a 24-hour glucose-fasting period to evaluate their need for basal insulin. Meals contain virtually no carbohydrates. Correcting doses of insulin are administered if preprandial glycemia is over 1.50 g/l or postprandial glycemia is over 2 g/l. Blood glucose levels must stay within normal values during the whole 24-hour period.
  Carbohydrate management is taught during meals and every afternoon through workshops about dietetics. Patients also learn how to deal with hypoglycaemia, hyperglycaemia and physical activity.
  A one-day follow-up takes place 3 months later.

SUMMARY:
The primary objective of this trial is to assess whether functional insulinotherapy decreases blood glucose variability at 3 months and 6 months, compared to initial values in type 1 diabetes patients.

So, this study measures the impact of functional insulinotherapy on several blood glucose variability indicators in patients with type 1 diabetes.

This trial also has a secondary objective: to measure the effect of functional insulinotherapy on oxidative stress and inflammation.

DETAILED DESCRIPTION:
This is a prospective, open, non-controlled study with an individual benefit for the participant. This study is designed to assess whether functional insulinotherapy decreases blood glucose variability at 3 months and 6 months, compared to initial values in type 1 diabetes patients.

All 30 patients with type 1 diabetes attended a 4-day functional insulinotherapy class, taught by 2 nurses, 2 dieticians and 2 physicians. The participants were recruited among metabolically stable patients who had already been prescribed functional insulinotherapy.

To assess the impact of functional insulinotherapy on blood glucose variability, HbA1c will be measured at 0, 3 months and 6 months along with 4 blood glucose variability indicators: MAGE, ADRR, LI and LBGI.

This trial also has a secondary objective: to measure the effect of functional insulinotherapy on oxidative stress. Therefore, a measure of insulin antibodies by ELISA at baseline. At baseline and 6 months, LTE4, TXB2, 8-iso-PGF2alpha, anti-transglutaminase and anti-endomysium antibodies will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes with pump or multi-injection treatment and attending a functional insulinotherapy class
* Social Security membership or benefit from Social Security
* Informed consent, with a signed and approved form

Exclusion Criteria:

* Underage patient, major patient under guardianship or protected by the Law
* Pregnant, parturient or breastfeeding woman
* Person with no freedom (prisoner), person in an emergency situation, person hospitalized without consent and not protected by the Law
* Antecedents of pathologies causing diabetes instability (coeliac disease, gastroparesis, non-balanced psychiatric pathology) and not optimally treated, acute pathology less than 3 months ago (infectious, cardio-vascular, metabolic), pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have been prescribed functional insulinotherapy at University Hospital Grenoble
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-09; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
MAGE, ADRR, Lability Index and LBGI computed with the blood glucose measurement or CGMS | 0, 3 months, 6 months

SECONDARY OUTCOMES:
anti-transglutaminase and anti-endomysium antibodies | 0 months, 6 months
dosage of urinary leucotriene E4 and 11-dehydro-thromboxane B2, 8-iso-PGF2alpha | 0 months, 6 months
anti-insulin antibodies by ELISA | 0 months

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Yves Benhamou, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Service de Diabétologie du Pr Halimi, CHU, Grenoble, France

REFERENCES:
- [Derived] Benhamou PY, Somers F, Lablanche S, Debaty I, Borel AL, Nasse L, Stanke-Labesque F, Faure P, Boizel R, Halimi S. Impact of flexible insulin therapy on blood glucose variability, oxidative stress and inflammation in type 1 diabetic patients: the VARIAFIT study. Diabetes Metab. 2014 Sep;40(4):278-83. doi: 10.1016/j.diabet.2014.01.004. Epub 2014 Feb 24. PMID 24581956